CLINICAL TRIAL: NCT04586764
Title: ST Elevation Myocardial Infarction Hemodynamic OutComes: Role of Non-Invasive Cardiac System (SHOCk-NICaS) Study
Acronym: SHOCk-NICaS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: University of Toronto (Other); University of British Columbia (Other); Scripps Health (Other); Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Ashish H Shah, Assistant Professor, University of Manitoba
Other Study IDs: HS22904
Record Dates: First submitted 2020-10-04; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: ST Elevation Myocardial Infarction (STEMI) Patients
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Non-Invasive Cardiac System — Non-Invasive Cardiac System (NICaS, NI Medical, Israel) is a non-invasive hemodynamic monitoring system that records various cardiovascular parameters including stroke volume, cardiac output, cardiac index (CI), total peripheral vascular resistance, body water content, and cardiac power index, a marker of myocardial contractility by employing the principles of the whole body impedance cardiography.

SUMMARY:
Proposed novel solution for high-risk heart disease Overall in-hospital mortality among ST elevation myocardial infarction (STEMI) patients is 3-4%, but >50% patients experiencing cardiogenic shock (CS) secondary to STEMI die in the hospital. Evidence suggests early diagnosis and treatment of CS results in improved outcomes, albeit, there is no tool to diagnose CS reliably in a timely fashion in STEMI patients through the continuous monitoring. We hypothesize that bioimpedance-derived hemodynamic measures obtained using the Non-Invasive Cardiac System (NICaS) can facilitate early detection of CS, predict outcomes, and revolutionize the STEMI patient management. The objectives of SHOCk-NICaS study in STEMI patients are to: a) identify the CS early, using NICaS derived cardiac index of ≤1.8L/min/m2 or ≤2.2L/min/m2 with the use of vasopressor and/or inotropes, and compare it with the incidence of CS based upon lactate level ≥2mmol/L, and systolic blood pressure <90mmHg; b): determine the impact of primary percutaneous coronary intervention (PPCI), using NICaS derived hemodynamic measures (stroke volume, cardiac index, cardiac power index, etc), by comparing pre- and post-angioplasty; and c) identify outcome-associated hemodynamic markers. A composite score of death during hospital stay, prolonged hospitalization due to heart failure (>72hrs), and use of inotropic or mechanical circulation support is a primary outcome.

Methodology This is a multi-center, double-blind, prospective cohort study enrolling STEMI patients aged ≥18years visiting at 4 cardiac centers (St Boniface, St. Michael's, McGill University Hospital). Using validated NICaS protocol, hemodynamic parameters will be recorded at baseline, during the PPCI procedure, and within 24-hour post PPCI without altering the standard care. Statistical analysis: Baseline data will be reported as mean±SD or median±interquartile range. The outcomes will be assessed using multivariable logistic regression. We will analyze the impact of age, sex, gender, and ethnicity on hemodynamic measures. The targeted 500 patients will ensure a margin of error of 5% at a 95% CI. So far recruited 76 STEMI patients mark the study feasibility.

Significance This novel study in high-risk STEMI patients will provide a promising cost-effective, rapid, and non-invasive tool to identify CS early; a prompt intervention may curtail the high morbidity and mortality. The meticulously designed pragmatic study outcomes may revolutionize STEMI patient management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years, presenting with EKG confirmed diagnosis of STEMI
* Able to understand, and consent to participate in the study

Exclusion Criteria:

* Patients unwilling to participate in the study
* Patients with any life-threatening medical condition with an expected life span of ≤1 year (e.g., metastatic cancer, terminal COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with STEMI
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Prolonged hospitalization due to heart failure (> 96 hours) | At 7 days
  Documented pulmonary edema on x-ray chest, elevated BNP or initiation of diuretic therapy lasting longer than 24 hours.
Use of inotropic - vasopressor therapy | At 7 days
  Use of norepinephrine, epinephrine, milrinone, dobutamine, or dopamine
Use of mechanical circulation support | At 7 days
  Intra aortic balloon pump, impella or extra-corporeal membrane oxygenation (ECMO) insertion
Death | At 7 days
Death | At 30 days
Death | At 1 year

SECONDARY OUTCOMES:
Killip classification | At 24 hours
  Killip class I - No signs of congestion Killip class II - Presence of S3 on clinical examination and/or basal rales on auscultation Class III - Acute pulmonary edema Class IV - Cardiogenic shock or hypotension (systolic blood pressure < 90 mmHg) and evidence of peripheral vasoconstriction characterized by oliguria, cold extremities or sweating.
New-onset atrial/ventricular arrhythmia | At 30 days
  Documented evidence of atrial - ventricular arrhythmia.
  Atrial fibrillation Atrial flutter Non-sustained ventricular tachycardia Sustained ventricular tachycardia Ventricular fibrillation
New-onset atrial/ventricular arrhythmia | From 30 days to 1 year
  Documented evidence of atrial - ventricular arrhythmia.
  Atrial fibrillation Atrial flutter Non-sustained ventricular tachycardia Sustained ventricular tachycardia Ventricular fibrillation
New diagnosis of heart failure | At 30 days
  Documented pulmonary edema on x-ray chest, elevated BNP or initiation of diuretic therapy lasting longer than 24 hours.
New diagnosis of heart failure | From 30 days to 1 year
  Documented pulmonary edema on x-ray chest, elevated BNP or initiation of diuretic therapy lasting longer than 24 hours.
Implantable Cardioverter Defibrillator (ICD) implantation | At 1 year
Cardiac Re-synchronization Therapy/Defibrillator (CRT-D) implantation | At 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet